CLINICAL TRIAL: NCT05432427
Title: 64Cu-DOTATATE PET-CT-skanning to Diagnose Macrophage Infiltration in the Heart Valves of Patients with Infective Endocarditis.
Brief Title: 64Cu-DOTATATE PET-CT-skanning and Infective Endocarditis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emil Loldrup Fosbol (Other)
Responsible Party: Sponsor-Investigator, Emil Loldrup Fosbol, Chief Physician, ph.d., Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-21040764
Record Dates: First submitted 2022-06-15; First posted 2022-06-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2022-06

CONDITIONS: Endocarditis; Endocarditis;Chronic; Endocarditis Acute
MeSH Terms: conditions — Endocarditis | interventions — 64Cu-DOTATATE; Fluorodeoxyglucose F18

STUDY DESIGN:
Intervention Model Description: Controlled prospectiv cohort study. Patients in the trial get a 64Cu-DOTATATEPET/ CT and/or 18F-FDG-PET/CT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group A, B, C, D, E, F, G (Experimental): Scans
  Interventions: Radiation: 64Cu-DOTATATE and 18F-FDG

INTERVENTIONS:
Radiation: 64Cu-DOTATATE and 18F-FDG — All participants will get a 64Cu-DOTATATE-PET and 18F-FDG-PET/CT.

SUMMARY:
The investigators hypothesize that the 64Cu-DOTATATE will show uptake in the infected vegetations on the prosthetic heart valves and increase the accuracy of the right diagnosis - thus increasing the sensitivity and specificity compared to 18F-FDG PET/CT

DETAILED DESCRIPTION:
Infective endocarditis (IE) is an infection of the heart lining, primarily mediated by an endothelial injury causing activation of inflammatory cytokines and cells thus forming a thrombus creating a basis for bacteria adherence. The incidence rate is estimated to 2-10 cases per 100.000 people. In hospital mortality rates have been reported to 14-30%. Hence,it is therefore also worrisome that the incidence of IE has significantly increased in the adult population the last decades. Several reasons for this incline in incidence have been suggested: an increasing elderly population, an increase in the prevalence of prosthetic heart valves and cardiac electronic devices and better diagnostics technique.

Prosthetic valve endocarditis (PVE) is uncommon but severe complication to surgical and transcatheter valve replacement. Early studies have estimated PVE to account for up to 5% of all IE cases, however in recent studies PVE represents an increased proportion of overall infective endocarditis cases -estimated for almost 20%. Staphylococcus aureus is the most common cause of PVE. The mortality rate of PVE patients is significantly higher than native valve endocarditis (NVE) - in hospital mortality is estimated from 22% to 42% for PVE, and one year mortality for PVE is estimated to 21%-80%. The PVE diagnosis is often hard to verify as the symptoms of IE vary broadly.18Fflurodeoxyglukocose positron emission tomography/computed tomography (18F-FDGPET/ CT) is recommended as diagnostic imaging technique, however the sensitivity is 83.5% and specificity is 70.8%. The aim of this trial is to investigate whether 64Cu-DOTATATE will show uptake in the infected vegetations on the prosthetic heart valves and increase the accuracy of the right diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Be able to understand given information and sign informered consent
* Group A: native heart valves without clinical or paraclinical sign of infection
* Group B: native heart valves with verified endocarditis (according to modified Duke-criteria)
* Group C: prothethic heart valves(mechanical or biological) without clinical or paraclinical sign of infection and more >1 year sind the heart operation
* Group D: infected prothethic heart valves, in addition clinical and paraclinical signs of infection (blood cultures and samples) and echocardiography
* Group E: newly operated in the heart valves without infection (6 months since operation)
* Group F: newly heart valve operation due to endocarditis (6 monts since operation)
* Group G: chronical infection in the aortic valce - lifelong antibiotics.

Exclusion Criteria:

* allergi for 64Cu-DOTATATE or 18-FDG
* obesity(weight over 140 kg)
* critically ill, and PET scan not possible
* Pregnancy or suspected pregnancy - negativ hCG will be required for fertile women
* severe claustrophobia
* diabetes - defined by farmacological treatment
* recent heart operation(<4 weeks)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-09-29 (Actual)

PRIMARY OUTCOMES:
The number(percentege) of agreement between the two scan modalities in overall population | 2 year
  x

SECONDARY OUTCOMES:
Compare the number of agreement in the uptake between the two scan modalities in infected patients versus newly operated patients | 2 year
  x

CONTACTS AND LOCATIONS:
Overall Officials: Emil L Fosbøl, MD,Ph.d., Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
The overall results of the trial